CLINICAL TRIAL: NCT01793337
Title: Tympanic and Frontal Versus Oesophageal Core Temperature Reading During Hot and Cold Environmental Exposure
Brief Title: Core Body Temperature Measurement During Hot and Cold Environmental Exposure
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institute of Mountain Emergency Medicine (Other)
Collaborators: Medical University Innsbruck (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Diagnostic
Other Study IDs: V/31/10
Record Dates: First submitted 2013-02-13; First posted 2013-02-15 (Estimated); Last update posted 2013-02-15 (Estimated); Status verified 2013-02

CONDITIONS: Body Temperature; Hypothermia
MeSH Terms: conditions — Hypothermia

ARMS (2):
- Cold first (Other): temperature is measured in cold (-20°C) environment first, and warm (23°C) environment afterwards
  Interventions: Other: Exposure to cold environmental temperature (-20°C)
- Warm first (Other): temperature is measured in warm (23°C) environment first, and cold (-20°C) environment afterwards
  Interventions: Other: Exposure to cold environmental temperature (-20°C)

INTERVENTIONS:
Other: Exposure to cold environmental temperature (-20°C)

SUMMARY:
Accurate measurement of core body temperature at the scene of an accident is critical for both diagnosis and treatment/triage decisions for hypothermic patients. Measurement in the lower third of the oesophagus is considered the gold standard of CT reading, but invasive and hardly applicable with a conscious patient. Tympanic membrane sensors for CT reading have been widely tested by may be unreliable in extreme environmental temperatures. Similarly, the Double Sensor device is a non-invasive device and is promising for prehospital use but has not been sufficiently verified under very cold and hot environmental conditions. Furthermore, comparisons of different non-invasive methods with oesophageal measurement in extreme conditions are lacking. The objective of these studies is to compare different techniques of core body temperature measurement with exposure to cold and hot environments.

ELIGIBILITY:
Inclusion Criteria:

* >18 years old
* ASA class 1

Exclusion Criteria:

* <18 years old
* American society of anesthesiologists class >1
* history of ear, nose, throat surgery
* congenital malformation of head/throat/ear/nose
* absence of informed consent

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2012-09; Primary Completion 2012-10 (Actual)

PRIMARY OUTCOMES:
Difference between oesophageal and epitympanic temperature | 10 min measurment at +20 °C followed by 10 min measurment at -20 °C

CONTACTS AND LOCATIONS:
Locations (1):
- Eurac research, Bolzano, Provincia autonoma di Bolzano, Italy

REFERENCES:
- [Background] Gunga HC, Werner A, Stahn A, Steinach M, Schlabs T, Koralewski E, Kunz D, Belavy DL, Felsenberg D, Sattler F, Koch J. The Double Sensor-A non-invasive device to continuously monitor core temperature in humans on earth and in space. Respir Physiol Neurobiol. 2009 Oct;169 Suppl 1:S63-8. doi: 10.1016/j.resp.2009.04.005. Epub 2009 Apr 14. PMID 19428314